CLINICAL TRIAL: NCT03479424
Title: Home Outpatient Monitoring and Engagement to Predict HF Exacerbation (HOME PREDICT-HF)
Brief Title: Home Outpatient Monitoring and Engagement to Predict HF Exacerbation
Acronym: Home Predict
Status: Terminated | Type: Observational
Why Stopped: Slow recruitment
Sponsor: University of California, San Francisco (Other)
Collaborators: MYIA Labs, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 18-24445
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: hospitalization
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training Set: n = 333
  Interventions: Other: Observational
- Validation Set: n = 167
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — The MYIA in-home suite of devices.
  Other Names: The MYIA in-home suite of devices.

SUMMARY:
The HOME PREDICT HF study looks at new ways to predict hospitalizations for heart failure. We will use a set of devices at home and surveys to collect information about patient's health. This study uses the Eureka app, a new study app developed by the University of California, San Francisco. The study is designed to happen remotely, using this application on a patient's smartphone, so that is as convenient as possible to participate.

DETAILED DESCRIPTION:
HOME PREDICT HF is single center, prospective, unblinded, randomly assigned training and validation observational cohorts to develop machine learning algorithms from an in-home suite of sensors in order to predict 3-month heart failure hospitalization and/or emergency department visits. Study population includes adults presenting with a diagnosis of reduced ejection fraction (LVEF <= 40%), NYHA class II-IV) who have had a hospitalization for HF in the previous 6 months. The study objectives include (1) To collect observational data from multiple sensors, patient-reported outcomes, and medical record data to develop (train) machine-learning algorithms (2) To validate trained algorithms in a separate validation cohort (3) To collect data to inform the design of a future intervention study. The primary outcome is Ninety-day heart failure hospitalization/emergency department visit for heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient and cared for by a PINNACLE Registry practice
2. Age ≥ 18 years old
3. Has a diagnosis of HF in the PINNACLE Registry/Medical Record
4. Seen by PINNACLE practice within the last 12 months
5. Has an LVEF ≤40% on their last data entry (within 1 year) in the PINNACLE Registry
6. NYHA Class II-IV by self-report
7. Has had a hospitalization for HF in the previous 6 months by self-report
8. Owns an Android or iOS smartphone, within Verizon cellular coverage zone in order to allow for data submission.
9. Sleep in the same bed at least 5 days per week
10. Willingness to complete the required surveys, measurements and study activities.

Exclusion Criteria:

1. Home oxygen use
2. Current or planned ventricular assist device
3. Previously or currently on a heart transplant list
4. Chronic dialysis
5. A diagnosis of any cancer and undergoing active treatment
6. In hospice or palliative care
7. Planned surgery/procedure in the next 3 months
8. Planned extended time away from home (>2 weeks) in the next 3 months
9. Living in a skilled nursing facility or other chronic care facility
10. Pregnancy or planned pregnancy in the next 3 months
11. Inability or unwillingness to consent and/or follow requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults presenting with a diagnosis of reduced ejection fraction (LVEF <= 40%), NYHA class II-IV) who have had a hospitalization for HF in the previous 6 months.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Heart Failure Hospitalization/ ED Visit | 90 day
  Ninety-day heart failure hospitalization/emergency department visit for heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Olgin, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No